CLINICAL TRIAL: NCT06435676
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of HRS9531 Tablets in Healthy Subjects
Brief Title: A Study of Single and Multiple Doses HRS9531 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-T-101
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Overweight or Obesity; Type 2 Diabetes
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD Stage: HRS9531 (Experimental): Administered po once
  Interventions: Drug: HRS9531
- SAD Stage: placebo (Placebo Comparator): Administered po once
  Interventions: Drug: Placebo
- MAD Stage: HRS9531 (Experimental): Administered po for multiple dose
  Interventions: Drug: HRS9531
- MAD Stage: placebo (Placebo Comparator): Administered po for multiple dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS9531 — Single dose escalation of HRS9531 tablets in healthy subjects
  Arms: SAD Stage: HRS9531
Drug: Placebo — Single dose of placebo in healthy adults
  Arms: SAD Stage: placebo
Drug: HRS9531 — Multiple dose escalation of HRS9531 tablets in healthy subjects
  Arms: MAD Stage: HRS9531
Drug: Placebo — Multiple dose of placebo in healthy adults
  Arms: MAD Stage: placebo

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of HRS9531tablets in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures, be able and willing to provide a written informed consent.
2. 18-55 years of age at the time of signing informed consent.
3. SAD stage: Body weight ≥50 kg,19.0 ≤BMI≤ 35.0 kg/m2 at screening visit. MAD stage: 24.0 ≤BMI≤ 35.0 kg/m2 at screening visit.
4. Subjects with good general health, no clinically significant abnormalities.

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial product(s) or related products.
2. With previous major organ diseases, including but not limited to neuropsychiatric, cardiovascular, digestive, respiratory, urinary, endocrine, blood, immune and other diseases, are judged by researchers to be unsuitable for the study.
3. Abnormal and clinically significant blood pressure at screening.
4. Blood donation within 1 month prior to screening, or blood donation ≥400 mL or blood loss ≥400 mL within 3 months prior to screening.
5. Participation in other clinical trials.
6. Presence of any clinically significant results in examination at screening visit.
7. Hepatitis B surface antigen (HBsAg), HIV antibody detection, treponema pallidum specific antibody detection, hepatitis C virus antibody (HCVAb) positive.
8. Presence of - clinically significant ECG results.
9. Known or suspected history of drug abuse or drug abuse, or urine drug screening test during the screening periodThose who are positive.
10. Addiction to tobacco and alcohol.
11. In the opinion of the investigator, there are any other conditions that interfere with the evaluation of the results of the trial or are not suitable for participation of this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
SAD Stage: Number of Adverse Events | 36 days
MAD Stage: Number of Adverse Events | 63 days

SECONDARY OUTCOMES:
Plasma Concentration-Time to Peak (Tmax) of HRS9531 | 36 days
  Tmax of a single dose of HRS9531 tablets
Area Under the Plasma Concentration-Time Curve (AUC) of HRS9531 | 36 days
  AUC of a single dose of HRS9531 tablets
Immunogenicity qualitative | 36 days
  anti-HRS9531 antibody
Plasma Concentration-Time to Peak (Tmax) of HRS9531 | 63 days
  Tmax of multiple dose of HRS9531 tablets
Area Under the Plasma Concentration-Time Curve (AUC) of HRS9531 | 63 days
  AUC of multiple dose of HRS9531 tablets
Glucose | 35 days
  fasting plasma glucose
Immunogenicity qualitative | 63 days
  anti-HRS9531 antibody

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital Of Anhui medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided